CLINICAL TRIAL: NCT03693534
Title: Clinical and Live Birth Rates After Controlled Ovarian Stimulation With the Long Antagonist Protocol Versus the Long Agonist Protocol
Brief Title: Clinical and Live Birth Rates After Following Long Antagonist Protocol Versus Long Agonist Protocol
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assisting Nature (Other)
Responsible Party: Principal Investigator, Papanikolaou Evaggelos, Papanikolaou Evaggelos, MD, PhD, Fertility Specialist, Scientific Director at Assisting Nature IVF Clinic, Assisting Nature
Other Study IDs: Long-Antagonist-AN005
Record Dates: First submitted 2018-09-24; First posted 2018-10-03 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Pregnancy, Ovarian
Keywords: Long Antagonist; Long agonist; clinical pregnancy rate; live birth rate; ovarian stimulation; IVF
MeSH Terms: conditions — Pregnancy, Ovarian

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Long Antagonist Protocol: Clinical Pregnancy Rate, Live Birth Rate and Blastulation Rate of patients who followed Long Antagonist Protocol for Controlled Ovarian Stimulation.
  Interventions: Diagnostic Test: Clinical Pregnancy Rate
- Long Agonist Protocol: Clinical Pregnancy Rate and Live Birth Rates and Blastulation Rate of patients who followed Long Agonist Protocol for Controlled Ovarian Stimulation.
  Interventions: Diagnostic Test: Clinical Pregnancy Rate

INTERVENTIONS:
Diagnostic Test: Clinical Pregnancy Rate — The Clinical Pregnancy, Live Birth Rate and Blastulation Rate according to the protocol of COS

SUMMARY:
A prospective study of the evaluation of the clinical IVF (in vitro fertilization) results after following Long Antagonist protocol for Controlled Ovarian Stimulation (COS) versus following Long Agonist protocol

DETAILED DESCRIPTION:
A prospective study of the clinical results in women who followed the Long Antagonist protocol for Controlled Ovarian Stimulation (COS) versus women who followed Long Agonist protocol, in an In Vitro Fertilization (IVF) try. In particular, the Clinical Pregnancy Rates (CPR) and Live Birth Rates (LBR) were estimated for the two groups of patients. The number of the formed blastocysts was also measured in each group of patients.

ELIGIBILITY:
Inclusion Criteria:

* primary infertility
* age 18-39 years; body mass index (BMI) 18-29kg/m2;
* regular menstrual cycle of 26-35days,
* presumed to be ovulatory;
* early follicular- phase serum concentration of FSH within normal limits (1-12 IU/l).

Exclusion Criteria:

* women with diabetes and other metabolic disease
* women with heart disease, QT prolongation,heart failure
* elevated liver enzymes, liver failure, hepatitis
* women with inflammatory or autoimmune disease
* abnormal karyotype;
* polycystic ovarian syndrome,
* endometriosis stage III/IV;
* history of being a 'poor responder',
* defined as >20 days of gonadotrophin in a previous stimulation cycle, or any previous cancellation of a stimulation cycle due to limited follicular response, or development of less than 4 follicles 15 mm in a previous stimulation cycle; history of recurrent miscarriage; severe OHSS in a previous stimula- tion cycle or any contraindication for the use of gonadotrophins.

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women 18- 39 years old who follow COS with the Long Antagonist Protocol or with Long Agonist Protocol
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2017-02-15 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Clinical Pregnancy Rate according to stimulation protocol | 6 weeks to 42 weeks after embryo transfer
  Clinical Pregnancy Rate according to stimulation protocol
Number of formed blastocysts in each group of patients | 5 days after the OPU day
  The number of the formed blastocysts in each group of patients according to the COS protocol

SECONDARY OUTCOMES:
Live Birth Rate according to stimulation protocol | 6 weeks to 42 weeks after embryo transfer
  Live Birth Rate according to stimulation protocol

CONTACTS AND LOCATIONS:
Overall Officials: Evaggelos Papanikolaou, MD, PhD, Principal Investigator — Assisting Nature; Robert Najdecki, MD, PhD, Principal Investigator — Assisting Nature
Locations (1):
- Assisting Nature, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: Undecided